CLINICAL TRIAL: NCT07238400
Title: Cardiac Effects of Mineralocorticoid Receptor Antagonism After Preeclampsia
Acronym: CARDAMOM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael C. Honigberg, Clinician Investigator, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P001799; R01HL181150 (NIH)
Record Dates: First submitted 2025-11-11; First posted 2025-11-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: Hypertension; Mineralocorticoid receptor; chlorthalidone; eplerenone; heart; microvascular; preeclampsia
MeSH Terms: conditions — Hypertension; Pre-Eclampsia | interventions — Eplerenone; Chlorthalidone; Potassium Chloride

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized, double-blind, active comparator clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eplerenone (Active Comparator): Participants will receive eplerenone 100 mg daily plus potassium placebo for 48 weeks
  Interventions: Drug: Eplerenone 100 mg daily; Drug: Potassium Placebo
- Chlorthalidone (Active Comparator): Participants will receive chlorthalidone 25 mg plus potassium 20 mEq daily for 48 weeks
  Interventions: Drug: Chlorthalidone 25 mg daily; Drug: Potassium Chloride

INTERVENTIONS:
Drug: Eplerenone 100 mg daily — Participants with a history of preeclampsia and current chronic hypertension will receive 100mg capsules of eplerenone to self-administer daily over the 48-week duration of the study treatment.
  Arms: Eplerenone
Drug: Chlorthalidone 25 mg daily — Participants with a history of preeclampsia with current chronic hypertension will receive 25mg capsules of chlorthalidone to self-administer daily over the 48-week duration of the study treatment.
  Arms: Chlorthalidone
Drug: Potassium Placebo — Participants taking eplerenone will also take a potassium placebo to self-administer daily over the 48-week duration of the study treatment.
  Arms: Eplerenone
Drug: Potassium Chloride — Participants taking chlorthalidone will also take 20 mEq of potassium to self-administer daily over the 48-week duration of the study treatment.
  Arms: Chlorthalidone

SUMMARY:
The goal of this clinical trial is to determine if the medication eplerenone yields greater improvements in coronary microvascular function than chlorthalidone in women who experienced preeclampsia during pregnancy and subsequently developed chronic hypertension. The main Aims are:

* To test the hypothesis that, in women with prior preeclampsia, current chronic hypertension, and concentric LV remodeling, eplerenone improves coronary microvascular function vs. chlorthalidone.
* To test the hypothesis that, in women with prior preeclampsia, current chronic hypertension, and concentric LV remodeling, eplerenone improves cardiac structure and function vs. chlorthalidone.

Participants will:

* First receive pre-treatment with Amlodipine for 12 weeks prior to beginning the study medication.
* Start study treatment which involves daily self-administration of two oral capsules (eplerenone + potassium placebo or chlorthalidone + potassium), each taken once a day, for a total of 336 doses over 48 weeks.
* Attend study visits at weeks 2, 12, 24, 36, and 48. These visits will involve collecting information, measuring blood pressure, and gathering blood and urine samples. Echocardiography (cardiac ultrasound), eye exam, and cardiac PET/CT scan will be performed during the baseline and week 48 visits.

DETAILED DESCRIPTION:
Preeclampsia, a condition marked by hypertension and systemic endothelial/microvascular dysfunction in late pregnancy, affects 8% of childbearing U.S. women and is associated with two-fold risk of future material cardiovascular disease (CVD). The American College of Cardiology and American Heart Association now recognize preeclampsia as a sex-specific CVD risk factor to guide prescription of preventive statin therapy. Beyond this focused recommendation, however, specific strategies for CVD risk reduction in women with preeclampsia are not yet established. Recent preclinical evidence suggests that preeclampsia induces vascular smooth muscle cell mineralocorticoid receptor (MR) sensitivity that persists postpartum, promoting hypertension and CVD. Although MR signaling is known to underlie hypertension, MR activation also promotes cardiovascular, kidney, and metabolic disease via effects that are partially independent of blood pressure. Work by this team has implicated MR signaling in coronary microvascular dysfunction, a known predictor of heart failure with preserved ejection fraction (HFpEF) and CVD mortality. The central hypothesis is that, among women with prior preeclampsia who subsequently develop chronic hypertension, MR blockade will promote favorable cardiac remodeling and improve coronary microvascular function, independent of changes in blood pressure, and thereby reduce CVD risk in affected women. To test this hypothesis, the investigators propose a randomized, double-blind clinical study in humans. Women aged <55 years with a history of preeclampsia, current chronic hypertension, and concentric left ventricular remodeling will be randomized 1:1 to receive eplerenone (mineralocorticoid receptor antagonist) or chlorthalidone (thiazide-like diuretic) with potassium supplementation for 48 weeks, targeting equivalent blood pressure control in both groups using daily home blood pressure measurement and 24-hour ambulatory blood pressure monitoring. The investigators will measure coronary microvascular function (myocardial flow reserve, i.e., hyperemic stress/rest myocardial blood flow) quantified by cardiac positron emission tomography (PET/CT) and cardiac structure and function by cardiac ultrasound at baseline and 48 weeks. It is expected that, compared with chlorthalidone, eplerenone will yield greater improvements in coronary microvascular function and myocardial diastolic function after 48 weeks of treatment. If the hypotheses are affirmed, these findings would support the targeted use of MR antagonists much earlier than recommended by current guidelines for the management of hypertension to more effectively prevent HFpEF and other CVD among women with a history of preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Female with a history of preeclampsia (defined by ACOG criteria) in a singleton pregnancy without pre-gestational chronic hypertension.
* Current chronic hypertension (stage 1 or greater).
* Evidence of concentric left ventricular (LV) remodeling, defined as relative LV wall thickness >0.42, with or without LV hypertrophy.
* Age 18-55 years at time of randomization.

Exclusion Criteria:

* Use of a mineralocorticoid receptor antagonist (MRA) or amiloride within the past 3 months or more than 30 days within the previous 12 months.
* Planned pregnancy, current pregnancy, or lactation.
* Systolic BP >150 mmHg and/or diastolic BP >95 mmHg while on antihypertensives, or systolic BP >160 mmHg and/or diastolic BP >100 mmHg if untreated.
* BMI >45 kg/m².
* Clinical atherosclerotic cardiovascular disease, including coronary, cerebrovascular, or peripheral artery disease.
* Diabetes mellitus.
* LV ejection fraction <40% or history of clinical heart failure (reduced or preserved ejection fraction).
* Hypertrophic or other genetic cardiomyopathy.
* Any moderate or greater valvular heart disease.
* eGFR <60 mL/min/1.73 m².
* Urine microalbumin/creatinine ratio >300 mg/g at screening.
* Abnormal electrolytes, hemoglobin, liver function tests, or TSH at screening or baseline.
* Plasma renin activity <1 mg/mL/hour and aldosterone >20 ng/dL (suggestive of primary aldosteronism).
* Use of oral contraceptives, progestin depot or implant (note: progestin-containing IUD is permitted), or menopausal hormone therapy.
* History of hypersensitivity or intolerance to calcium channel blockers, thiazides, or MRAs.
* Active substance abuse.
* Other serious medical illnesses or concerns about protocol adherence/mortality risk within 15 months.
* Participation in another interventional clinical study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-03-16 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Myocardial Flow Reserve (MFR) | Prior to randomization and after 48 weeks of randomized study treatment.
  Subjects will undergo 13N cardiac PET imaging at baseline and after 48 weeks of randomized study treatment. Myocardial blood flow (MBF) will be determined during the stress and rest conditions. Myocardial flow reserve will be calculated as stress MBF divided by rest MBF.

SECONDARY OUTCOMES:
Ratio of mitral E velocity to e' [E/e'] | Prior to randomization and after 48 weeks of randomized study treatment.
  E/e', a measure of diastolic function, will be measured by transthoracic echocardiography.
Rest Myocardial Blood Flow (MBF) | Prior to randomization and after 48 weeks of randomized study treatment.
  Subjects will undergo 13N cardiac PET imaging at baseline and after 48 weeks of randomized study treatment. Myocardial blood flow (MBF) will be determined during the stress and rest conditions.
Stress Myocardial Blood Flow (MBF) | Prior to randomization and after 48 weeks of randomized study treatment.
  Subjects will undergo 13N cardiac PET imaging at baseline and after 48 weeks of randomized study treatment. Myocardial blood flow (MBF) will be determined during the stress and rest conditions.
Subendocardial-Specific Myocardial Flow Reserve (MFR) | Prior to randomization and after 48 weeks of randomized study treatment.
  Subjects will undergo 13N cardiac PET imaging at baseline and after 48 weeks of randomized study treatment. Myocardial blood flow (MBF) will be determined during the stress and rest conditions. Subendocardial layer-specific MBF will be calculated using QPET software (Cedars-Sinai Medical Center, Los Angeles, CA). Myocardial flow reserve will be calculated as stress MBF divided by rest MBF.
Relative wall thickness | Prior to randomization and after 48 weeks of randomized study treatment.
  Relative wall thickness is calculated as 2*posterior wall thickness/LV end-diastolic diameter as measured by transthoracic echocardiography.
Early diastolic septal mitral annular velocity [septal e'] | Prior to randomization and after 48 weeks of randomized study treatment.
  Septal e', a measure of diastolic function, will be measured by transthoracic echocardiography using tissue Doppler.
Peak tricuspid regurgitant velocity | Prior to randomization and after 48 weeks of randomized study treatment.
  Peak tricuspid regurgitant jet velocity, a measure of diastolic function, will be measured by transthoracic echocardiography using continuous wave Doppler.
Left atrial volume index | Prior to randomization and after 48 weeks of randomized study treatment.
  Left atrial volume index will be measured by transthoracic echocardiogarphy using the biplane method and indexed for body surface area.
Left atrial reservoir strain | Prior to randomization and after 48 weeks of randomized study treatment.
  Left atrial strain, a sensitive measure of end-diastolic pressure and atrial remodeling, will be quantified using TOMTEC.
Peak global longitudinal strain | Prior to randomization and after 48 weeks of randomized study treatment.
  Left ventricular global longitudinal strain, a measure of subclinical cardiac dysfunction, will be quantified using TOMTEC.

OTHER OUTCOMES:
Renal blood flow | Prior to randomization and after 48 weeks of randomized study treatment.
  Renal blood flow is calculated from 13N cardiac PET images. Rest and stress renal blood flow are estimated by fitting the tissue time-activity curves to a 2-compartment kinetic model.
Retinal vessel density | Prior to randomization and after 48 weeks of randomized study treatment.
  For OCT ocular retinal imaging, subjects will be scanned on the commercially available spectral domain OCT machine (AngioVue OCTA, RTVue, Optovue Inc., Fremont, CA). Ocular imaging will include the 3 main retinal parameters available with the latest software package: (1) foveal avascular zone size, (2) peripapillary vessel density and internal limiting membrane-nerve fiber layer thickness, and (3) macular vessel density and macular internal limiting membrane-inner plexiform layer thickness and macular internal limiting membrane-retinal pigment epithelium full retinal thickness.
Concentration of High-sensitivity cardiac troponin I | Prior to randomization and after 48 weeks of randomized study treatment.
  High-sensitivity cardiac troponin I, a marker of cardiovascular injury and remodeling, will be measured via blood collection.
Level of N-terminal pro-B-type natriuretic peptide | Prior to randomization and after 48 weeks of randomized study treatment.
  NT-proBNP, a marker of cardiac wall stretch and remodeling, will be measured via blood collection.
High-sensitivity C-reactive protein | Prior to randomization and after 48 weeks of randomized study treatment.
  We will measure high-sensitivity C-reactive protein, a marker of inflammation and cardiovascular disease risk, via blood collection.
Level of Interleukin-6 | Prior to randomization and after 48 weeks of randomized study treatment.
  IL-6, a marker of inflammation and cardiovascular disease risk, will be measured via blood collection.
Concentration of Transforming growth factor-beta1 | Prior to randomization and after 48 weeks of randomized study treatment.
  TGF-B1, a marker of fibrosis, will be measured via blood collection.
Concentration of procollagen type I carboxy-terminal propeptide | Prior to randomization and after 48 weeks of randomized study treatment.
  PICP, a marker of fibrosis, will be measured via blood collection.
Urine microalbumin-to-creatinine ratio | Prior to randomization and after 48 weeks of randomized study treatment.
  Microalbumin-to-creatinine will be measured through urine.
Score of Coronary artery calcium | Prior to randomization and after 48 weeks of randomized study treatment.
  Gated CT will be performed with cardiac PET scans. Coronary artery calcium scores will be quantified using the Agatston method and can range from 0 (no plaque) to more than 1000 (extensive plaque).
24-hour ambulatory blood pressure | Prior to randomization and after 48 weeks of randomized study treatment.
  24-hour BP monitoring will be performed as part of the baseline and post-treatment assessments using a validated ambulatory BP monitor (WatchBP O3, microlife, Clearwater, FL). Mean 24- hour systolic and diastolic BP will be calculated from the device data.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Honigberg, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No